CLINICAL TRIAL: NCT02549911
Title: Hyperthermic Intraperitoneal Chemotherapy, Intravenous Chemotherapy Combined With Surgery for the Treatment of Advanced Gastric Cancer With Peritoneal Metastasis
Brief Title: HIPEC, Intravenous Chemotherapy and Surgery for the Treatment of Advanced GC With Peritoneal Metastasis
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhejiang Cancer Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HISA
Record Dates: First submitted 2015-09-07; First posted 2015-09-15 (Estimated); Last update posted 2015-09-15 (Estimated); Status verified 2015-09

CONDITIONS: Gastric Cancer
Keywords: chemotherapy; surgery; Surgically-Created Resection Cavity; Adverse Reaction to Drug
MeSH Terms: conditions — Stomach Neoplasms; Drug-Related Side Effects and Adverse Reactions | interventions — Hyperthermic Intraperitoneal Chemotherapy; Drug Therapy; Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- HIPEC,Chemotherapy AND surgery (Experimental): 1. surgical exploration,if PCI<20,then we perform this study
  2. HIPEC（RHL-2000B, Madain Medical Devices Co., Ltd., Jilin, China): Taxol (Paclitaxel Injection) 75 mg/m2, twice, within 72 hours after surgical exploration ; oral chemotherapy:S-1(Tegafur,Gimeracil and Oteracil Potassium Capsules): 80mg/m2, twice daily (after the breakfast and supper) for two weeks, and then suspend for one week.
  3. chemotherapy(3 cycles) : Taxol 150mg/m2,d1, S-1: 80mg/m2, twice daily (after the breakfast and supper) for two weeks, and then suspend for one week.
  4. surgery:Secondary surgical exploration:if PCI less than 20,then perform the cytoreductive surgery(resection of primary tumors and metastases )
  5. after the surgery,HIPEC for two cycles,and PS chemotherapy for 3 cycles
  Interventions: Other: HIPEC,Chemotherapy AND surgery

INTERVENTIONS:
Other: HIPEC,Chemotherapy AND surgery — 1. HIPEC（RHL-2000B, Madain Medical Devices Co., Ltd., Jilin, China): Taxol (Paclitaxel Injection) 75 mg/m2, twice, within 72 hours after surgical exploration ; oral chemotherapy:S-1(Tegafur,Gimeracil and Oteracil Potassium Capsules): 80mg/m2, twice daily (after the breakfast and supper) for two weeks, and then suspend for one week.
  2. chemotherapy(PS for 3 cycles) : Taxol 150mg/m2,d1, S-1: 80mg/m2, twice daily (after the breakfast and supper) for two weeks, and then suspend for one week.
  3. surgery:Secondary surgical exploration:if PCI less than 20,then perform the cytoreductive surgery(resection of primary tumors and metastases )
  4. after the surgery,HIPEC for two cycles,and PS chemotherapy for 3 cycles

SUMMARY:
Explore the hyperthermic intraperitoneal chemotherapy (HIPEC) and intravenous chemotherapy for Creating the Operation Chance in advanced gastric cancer with peritoneal metastasis.

DETAILED DESCRIPTION:
To assess the effectiveness and safety of Hyperthermic intraperitoneal chemotherapy, intravenous chemotherapy combined with surgery for the treatment of advanced gastric cancer with peritoneal metastasis,so as to further find out the optimal protocol for the Conversion therapy in the patients with advanced gastric cancer.

ELIGIBILITY:
Inclusion Criteria:

gastric cancer confirmed by endoscopic biopsy , and enhanced CT suspected to have peritoneal metastasis, including ascites, ovarian metastasis, omentum or peritoneal metastasis.

* Definitely diagnosed as above stage of stomach cancer before the operation via CT or MRI, ultrasonic endoscopy and blood tumor antigen test, or through the laparoscopy if necessary
* Untreated (e.g. radiotherapy, chemotherapy, target therapy and immunotherapy)
* ECOG (Eastern Cooperative Oncology Group) : 0~2
* Age: 18~75 years old
* Normal hemodynamic indices before the recruitment (including blood cell count and liver/kidney function). For example: WBC>4.0×109/L, NEU >1.5×109/L, PLT>100×109/L, BIL<1.5 times of upper limit of normal reference value, ALT and AST<2.5 times of upper limit of normal reference value, and CRE<1.2mg/dl
* Good cardiac function before the recruitment, no seizure of myocardial infarction in past half year, and controllable hypertension and other coronary heart diseases
* Not concomitant with other uncontrollable benign diseases before the recruitment (e.g. the infection in the lung, kidney and liver)
* Not participating in other study projects before and during the treatment
* Signed the Informed Consent Form

Exclusion Criteria:

* Not conforming to above inclusion criteria
* Distal metastasis to lung, liver, or para aortic lymph node metastasis
* Ever operation on the stomach
* Operation intolerance due to other systemic basic diseases
* Ever administered other drugs (including TCM drugs) before the recruitment, or no guarantee of progress according to the study requirement after the recruitment
* Allergy to the drugs in this protocol
* Pregnant or lactating women
* Women at childbearing age and of pregnancy desire during the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2015-09; Primary Completion 2016-09 (Estimated); Study Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
R0 resection | 3 months
  the rate of R0 resection

SECONDARY OUTCOMES:
Adverse Events | 6 months
  Number and degree of Adverse Events
Overall survival time | 3 years
  the overall survival time

CONTACTS AND LOCATIONS:
Overall Officials: Yian Du, MD, Principal Investigator — Zhejiang Cancer Hospital
Locations (1):
- Zhejiang Cancer Hospital, Hangzhou, Zhejiang, China

REFERENCES:
- [Background] Wu X, Li Z, Li Z, Jia Y, Shan F, Ji X, Bu Z, Zhang L, Wu A, Ji J. Hyperthermic intraperitoneal chemotherapy plus simultaneous versus staged cytoreductive surgery for gastric cancer with occult peritoneal metastasis. J Surg Oncol. 2015 Jun;111(7):840-7. doi: 10.1002/jso.23889. Epub 2015 Apr 10. PMID 25864884
- [Background] Xia W, Hu Y, Mou T, Chen T, Yu J, Li G. [Safety and efficacy of intraperitoneal hyperthermic perfusion chemotherapy following laparoscopic palliative resection for gastric cancer patients with peritoneal metastasis]. Zhonghua Wei Chang Wai Ke Za Zhi. 2014 Nov;17(11):1087-91. Chinese. PMID 25421766
- [Background] Di Vita M, Cappellani A, Piccolo G, Zanghi A, Cavallaro A, Bertola G, Bolognese A, Facchini G, D'Aniello C, Di Francia R, Cardi F, Berretta M. The role of HIPEC in the treatment of peritoneal carcinomatosis from gastric cancer: between lights and shadows. Anticancer Drugs. 2015 Feb;26(2):123-38. doi: 10.1097/CAD.0000000000000179. PMID 25406023
- [Derived] Yu P, Ye Z, Dai G, Zhang Y, Huang L, Du Y, Cheng X. Neoadjuvant systemic and hyperthermic intraperitoneal chemotherapy combined with cytoreductive surgery for gastric cancer patients with limited peritoneal metastasis: a prospective cohort study. BMC Cancer. 2020 Nov 16;20(1):1108. doi: 10.1186/s12885-020-07601-x. PMID 33198674